CLINICAL TRIAL: NCT01496989
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate Safety and Immunogenicity of a Multiantigen HIV (HIV-MAG) pDNA Vaccine With or Without Human IL-12 pDNA GENEVAX® IL-12) and Ad35-GRIN/ENV Vaccine in HIV-Uninfected, Healthy Volunteers
Brief Title: Safety and Immunogenicity Study of HIV-MAG Vaccine +/- IL-12 and Ad35-GRIN/ENV in HIV-uninfected Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Auro Vaccines LLC (Industry); Ichor Medical Systems Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI B004
Record Dates: First submitted 2011-12-19; First posted 2011-12-22 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; HIV vaccine; HIV prevention
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1: HIV-MAG followed by Ad35-GRIN/ENV (Experimental): HIV-MAG (IM/EP) at Months 0,1,2 followed by Ad35-GRIN/ENV (IM) at Month 6. (Vaccine:Placebo = 12/3)
  Interventions: Biological: HIV-MAG (3,000mcg); Biological: Ad35-GRIN/ENV
- Group 2: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV (Experimental): HIV-MAG + GENEVAX® IL-12 (IM/EP) at Months 0,1,2 followed by Ad35-GRIN/ENV (IM) at Month 6. (Vaccine:Placebo=12/3)
  Interventions: Biological: HIV-MAG (3,000mcg); Biological: GENEVAX® IL-12 (100mcg); Biological: Ad35-GRIN/ENV
- Group 3: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV (Experimental): HIV-MAG + GENEVAX® IL-12 (IM/EP) at Months 0,1,2 followed by Ad35-GRIN/ENV (IM) at Month 6. (Vaccine:Placebo= 12/3)
  Interventions: Biological: HIV-MAG (3,000mcg); Biological: GENEVAX® IL-12 (1000mcg); Biological: Ad35-GRIN/ENV
- Group 4: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV (Experimental): HIV-MAG + GENEVAX® IL-12 (IM/EP) at Month 0 followed by Ad35-GRIN/ENV (IM) at Month 4. (Vaccine:Placebo=12/3)
  Interventions: Biological: HIV-MAG (3,000mcg); Biological: GENEVAX® IL-12 (1000mcg); Biological: Ad35-GRIN/ENV
- Group 5: Ad35-GRIN/ENV followed by HIV-MAG+GENEVAX® IL-12 (Experimental): Ad35-GRIN/ENV (IM) at Month 0 followed by HIV-MAG + GENEVAX® IL-12 (IM/EP) at Month 4. (Vaccine:Placebo=12/3)
  Interventions: Biological: HIV-MAG (3,000mcg); Biological: GENEVAX® IL-12 (1000mcg); Biological: Ad35-GRIN/ENV

INTERVENTIONS:
Biological: HIV-MAG (3,000mcg) — Delivered intramuscularly by in vivo electroporation
Biological: GENEVAX® IL-12 (100mcg) — Co-administered with HIV-MAG, delivered intramuscularly by in vivo electroporation
  Arms: Group 2: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV
Biological: GENEVAX® IL-12 (1000mcg) — Co-administered with HIV-MAG, delivered intramuscular by in vivo electroporation
  Arms: Group 3: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV; Group 4: HIV-MAG+GENEVAX® IL-12 followed by Ad35-GRIN/ENV; Group 5: Ad35-GRIN/ENV followed by HIV-MAG+GENEVAX® IL-12
Biological: Ad35-GRIN/ENV — (2x10^10vp) Delivered intramuscularly by standard needle injection

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and immunogenicity of multiantigen HIV (HIV-MAG) plasmid DNA (pDNA) vaccine co-administered with recombinant human IL-12 pDNA (GENEVAX® IL-12) followed or preceded by recombinant Ad35-GRIN/ENV HIV vaccine in low-risk for HIV-uninfected healthy adults.

DETAILED DESCRIPTION:
The study is a randomized, double-blind placebo-controlled trial assessing the safety and tolerability of HIV-MAG with or without co-administered GENEVAX® IL-12 given intramuscularly by in vivo electroporation (IM/EP) using the Ichor Medical Systems TriGrid Delivery System (TDS-IM) followed by Ad35-GRIN/ENV in each of four different regimens. An additional group will evaluate the safety and tolerability of Ad35-GRIN/ENV followed by HIV-MAG with co-administered GENEVAX® IL-12 given intramuscularly by in vivo electroporation (IM/EP) using the Ichor Medical Systems TriGrid Delivery System (TDS-IM).

Volunteers will be screened up to 42 days before the 1st vaccination and will be followed for 12 months after the first vaccine administration. It is anticipated that it will take approximately 3 months to enrol the study. Approximately 75 volunteers (60 vaccine/15 placebo recipients) will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female adults,
* 18 to 50 years of age (21 to 50 years of age for volunteers in Rwanda),
* who do not report high-risk behaviour for HIV infection,
* who are available for the duration of the trial,
* who are willing to undergo HIV testing,
* use an effective method of contraception, and
* who, in the opinion of the principal investigator or designee, understand the study and who provide written informed consent.

Principal exclusion criteria:

* confirmed HIV infection,
* pregnancy and lactation,
* significant acute or chronic disease,
* clinically significant laboratory abnormalities,
* recent vaccination or receipt of a blood product,
* previous receipt of an HIV vaccine, and
* previous severe local or systemic reactions to vaccination or history of severe allergic reactions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 13 months approximately
  To evaluate the safety and tolerability of HIV-MAG, GENEVAX® IL-12, and Ad35-GRIN/ENV administered in five heterologous prime-boost regimens.

SECONDARY OUTCOMES:
Immunogenicity | 12 months
  To assess (qualitative and quantitative) immune responses elicited by the different prime-boost regimens.

CONTACTS AND LOCATIONS:
Locations (3):
- Kenya AIDS Vaccine Initiative, Kangemi, Nairobi, Kenya
- Projet San Francisco, Kigali, Rwanda
- Uganda Virus Research Institute-IAVI, Entebbe, Uganda

REFERENCES:
- [Derived] Mpendo J, Mutua G, Nanvubya A, Anzala O, Nyombayire J, Karita E, Dally L, Hannaman D, Price M, Fast PE, Priddy F, Gelderblom HC, Hills NK. Acceptability and tolerability of repeated intramuscular electroporation of Multi-antigenic HIV (HIVMAG) DNA vaccine among healthy African participants in a phase 1 randomized controlled trial. PLoS One. 2020 May 29;15(5):e0233151. doi: 10.1371/journal.pone.0233151. eCollection 2020. PMID 32469893
- [Derived] Mpendo J, Mutua G, Nyombayire J, Ingabire R, Nanvubya A, Anzala O, Karita E, Hayes P, Kopycinski J, Dally L, Hannaman D, Egan MA, Eldridge JH, Syvertsen K, Lehrman J, Rasmussen B, Gilmour J, Cox JH, Fast PE, Schmidt C. A Phase I Double Blind, Placebo-Controlled, Randomized Study of the Safety and Immunogenicity of Electroporated HIV DNA with or without Interleukin 12 in Prime-Boost Combinations with an Ad35 HIV Vaccine in Healthy HIV-Seronegative African Adults. PLoS One. 2015 Aug 7;10(8):e0134287. doi: 10.1371/journal.pone.0134287. eCollection 2015. PMID 26252526
- See also: International AIDS Vaccine Initiative — http://www.iavi.org
- See also: Ichor Medical Systems, Inc. — http://www.ichorms.com/